CLINICAL TRIAL: NCT01882413
Title: A Study to Determine the Prevalence of Inflammatory Dry Eye Disease in Patients Prior to Cataract Removal
Acronym: REVEAL
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-RES-012-001
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Planned Cataract Removal: Patients with planned cataract removal surgery are evaluated for the presence of inflammatory dry eye disease. No treatment is administered.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study will evaluate the prevalence of inflammatory dry eye disease in patients prior to cataract surgery. No treatment is administered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo cataract removal surgery

Exclusion Criteria:

* Current use of eye drops or oral medications for allergic conjunctivitis
* Serious ocular injury, intraocular surgery, or refractive surgery within 6 months in the study eye
* Use of a contact lens within 4 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with planned cataract removal surgery
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (6):
- Canada (6):
  - Brandon, Manitoba
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Boisbriand, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Planned Cataract Removal
Started | 204
Completed | 204
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Presence of Matrix Metalloproteinase-9 (MMP-9) in the Study Eye
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye.
Time Frame: Up to 60 Days Prior to Surgery
Population: Per-protocol population included all enrolled participants who completed all the study assessments without major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 199
percentage of participants | 36.2

2. Secondary Outcome: Percentage of Participants Suspected of Having Dry Eye With Elevated MMP-9
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. Suspected of having dry eye was defined as a response of "Yes" to the Investigator Dry Eye History question.
Time Frame: Up to 60 days prior to cataract surgery
Population: Participants from the Per-protocol population, all enrolled participants who completed all the study assessments without major protocol violations, with elevated data MMP-9 and data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 39
percentage of participants | 23.1

3. Secondary Outcome: Percentage of Participants With Elevated MMP-9 Without Prior Diagnosis or Physician Recommended Intervention
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. Participants without a prior diagnosis of keratoconjunctivitis sicca, dry eye or tear film insufficiency or physician recommended use of topical cyclosporine, artificial tears or punctal plugs are included in the analysis.
Time Frame: Up to 60 days prior to cataract surgery
Population: Participants from the Per-protocol population, all enrolled participants who completed all the study assessments without major protocol violations, with elevated MMP-9 and data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 142
percentage of participants | 36.6

4. Secondary Outcome: Percentage of Participants With Elevated MMP-9 With Dry Eye Symptoms Without Conjunctival or Corneal Staining
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. Dry eye symptoms were measured by a score of at least ≥ 2 using the Subject Evaluation of Symptoms of Dryness (SESoD) questionnaire without conjunctival or corneal staining. The SESoD assesses dry eye using a 5-point scale where 0= no dryness to 4= severe dryness. Conjunctival and Corneal Staining were evaluated as part of the slit lamp biomicroscopy examination. Eye structures and surfaces were assessed for dry eye signs using a 5-point scale where: 0=none, 0.5=trace, 1=mild, 2=moderate and 3=severe. Higher values represent a worse outcome.
Time Frame: Up to 60 days prior to cataract surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 16
percentage of participants | 12.5

5. Secondary Outcome: Percentage of Participants With Elevated MMP-9 With Dry Eye Symptoms Without Any Signs
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. Dry eye symptoms were measured by a score of at least ≥ 2 using the SESoD questionnaire without any signs. The SESoD assesses dry eye using a 5-point scale where 0= no dryness to 4= severe dryness. Signs included conjunctival or corneal staining, Schirmer's score ≤ 7mm, or Tear Film Break-up Time [TFBUT] ≤ 10 seconds.
Time Frame: Up to 60 days prior to cataract surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 3
percentage of participants | 33.3

6. Secondary Outcome: Percentage of Participants With Elevated MMP-9 With at Least One Dry Eye Sign Without Dry Eye Symptoms
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. Dry Eye Signs included conjunctival or corneal staining, Schirmer's score ≤ 7 mm, or Tear Film Break-up Time [TFBUT] ≤ 10 seconds without Dry eye symptoms measured by a score of at least ≤ 1 using the SESoD questionnaire. The SESoD assessed dry eye using a 5-point scale where 0= no dryness to 4= severe dryness.
Time Frame: Up to 60 days prior to cataract surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 131
percentage of participants | 38.2

7. Secondary Outcome: Percentage of Participants With Elevated MMP-9 With at Least One Dry Eye Sign and Dry Eye Symptoms
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. Dry Eye Signs included conjunctival or corneal staining, Schirmer's score ≤ 7mm, or Tear Film Break-up Time [TFBUT] ≤ 10 seconds with Dry eye symptoms measured by a score of at least ≥ 2 using the SESoD questionnaire. The SESoD assessed dry eye using a 5-point scale where 0= no dryness to 4= severe dryness.
Time Frame: Up to 60 days prior to cataract surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 58
percentage of participants | 29.3

8. Secondary Outcome: Percentage of Participants With Elevated MMP-9 Who Routinely Use Artificial Tears
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. Artificial Tear usage was assessed by the investigator.
Time Frame: Up to 60 Days Prior to Surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 49
percentage of participants | 34.7

9. Secondary Outcome: Percentage of Participants With Elevated MMP-9 With Punctal Plugs
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. A history of punctual plug usage was assessed by the investigator.
Time Frame: Up to 60 Days Prior to Surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 1
percentage of participants | 0

10. Secondary Outcome: Percentage of Participants With Elevated MMP-9 With Corneal Staining Grade ≥ 1 and ≥ 2
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. Corneal Staining was evaluated as part of the slit lamp biomicroscopy examination. Eye structures and surfaces were assessed for signs of dry eye using a 5-point scale where: 0=none, 0.5=trace, 1=mild, 2=moderate and 3=severe. Higher values represent a worse outcome.
Time Frame: Up to 60 Days Prior to Surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 105
percentage of participants
  Grade ≥ 1 | 37.1
  Grade ≥ 2 (n=43) | 41.9

11. Secondary Outcome: Percentage of Participants With Elevated MMP-9 and an Ocular Surface Disease Index® (OSDI®) > 12, > 22 and ≥ 32
Description: Tear film was collected and a diagnostic test was used to determine the presence of MMP-9 in the study eye. The OSDI consists of 12 questions to assess visual function, ocular symptoms and environmental triggers related to dry eye. Each of the 12 questions is assessed using a 5-point scale (0=none of the time to 4=all of the time) which is converted to a total score between 0-100. OSDI total scores of 0-12=normal (best), 13-22= mild ocular surface disease, 23-32 =moderate ocular surface disease, and 33-100=severe ocular surface disease (worst).
Time Frame: Up to 60 Days Prior to Surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Planned Cataract Removal
Number analyzed (Participants) | 199
percentage of participants
  OSDI > 12 (n=116) | 39.7
  OSDI > 22 (n=76) | 46.1
  OSDI > 32 (n=50) | 46.0

ADVERSE EVENTS:
Time Frame: Adverse Events that did not resolve by the end of Baseline Visit 1 were followed for up to 30 days.
Arm/Group | Patients With Planned Cataract Removal
Serious Adverse Events (participants affected / at risk) | 0/204
Other Adverse Events (participants affected / at risk) | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.